CLINICAL TRIAL: NCT06544720
Title: A Phase 1 Clinical Study of Autologous TCR-T Cells (SCG142) Therapy for Advanced HPV Associated Carcinomas
Brief Title: SCG142 TCR-T Cells for Human Papillomavirus-Associated Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCG142-CI-101
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Human Papillomavirus Associated Carcinomas; Cervical Cancer; Head and Neck Cancers; Anal Cancer; Vulva Cancer; Vaginal Cancer; Penile Cancer; HPV-Related Malignancy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Head and Neck Neoplasms; Anus Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Penile Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCG142 TCR-T cells (Experimental): Monotherapy of SCG142
  Interventions: Biological: SCG142 TCR-T cells

INTERVENTIONS:
Biological: SCG142 TCR-T cells — Monotherapy of SCG142

SUMMARY:
A multicenter, open, single arm dose escalation and dose expansion phase I study to evaluate the safety, tolerability, and efficacy of SCG142 TCR-T cells in Subjects with advanced HPV associated carcinomas.

ELIGIBILITY:
Key Inclusion Criteria:

1. Greater than or equal to 18 years of age
2. HPV associated carcinomas
3. Patients must have at least one measurable lesion defined by RECIST 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Key Exclusion Criteria:

1. Active or uncontrollable infections or other active major medical illnesses of the cardiovascular, respiratory.
2. Patients with active autoimmune diseases.
3. Patient has a known active Hepatitis B or Hepatitis C.
4. Other severe medical conditions that may limit subject's participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT | 28 days
  Number of subjects with adverse events (AEs) and laboratory abnormalities defined as dose limiting toxicities (DLT)

SECONDARY OUTCOMES:
Efficacy: antitumor activity of SCG142 | 2 years
  Assessed by RECIST 1.1 and iRECIST

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hosptial of qingdao university, Qingdao, Shandong, China